CLINICAL TRIAL: NCT05430269
Title: Faecal Bacteriotherapy for Antibiotic-Associated Diarrhoea in Patients In Intensive Care - Randomised Controlled Trial
Brief Title: Faecal Bacteriotherapy for Postantibiotic Diarrhoea in Critically Ill Patients
Acronym: FEBATRICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Faculty Hospital Kralovske Vinohrady (Other Government); Donatio Intensivistam Endowment Fund (Unknown)
Responsible Party: Principal Investigator, Frantisek Duska, MD, PhD, František Duška, MD, PhD, A/Prof, AFICM, EDIC, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-002290-25
Record Dates: First submitted 2022-04-03; First posted 2022-06-24 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Diarrhea Caused by Drug; Clostridium Difficile Infections
Keywords: gut microbiota; critically ill; fecal microbial transplantation
MeSH Terms: conditions — Clostridium Infections; Critical Illness | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Prospective, single center, parallel group randomised controlled trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): ICU patients who developed diarhea after a course of antibiotic therapy treated with Faecal bacteriotherapy (FBT) delivered as enema
  Interventions: Other: Faecal bacteriotherapy (FBT)
- Control group (Active Comparator): ICU patients who developed diarhea after a course of antibiotic therapy treated standard-of-care protocolised treatment of postantibiotic diarhea
  Interventions: Other: standard-of-care protocolised treatment of postantibiotic diarhea

INTERVENTIONS:
Other: Faecal bacteriotherapy (FBT) — Enema of 350 ml of standardised mixed transplantate prepared from faeces of 7 healthy donors.
  Arms: Intervention group
Other: standard-of-care protocolised treatment of postantibiotic diarhea — standard-of-care protocolised treatment of postantibiotic diarhea
  Arms: Control group

SUMMARY:
Rationale: Postantibiotic diarrhoea in critically ill patients is common, often prolonged and currently there is no effective treatment of it.

Aim: To test safety and feasibility of faecal microbial transplantation in critically ill patients with postantibiotic diarhoea.

Design: Prospective, single center, parallel group randomised controlled trial. Subjects: ICU patients (both general and burn ICU) who developed diarhea after a course of antibiotic therapy that is persistent for 24 hours and is not due to other causes. Patients with septic shock or approaching death will be excluded.

Treatment in the intervention group: Faecal bacteriotherapy (FBT) delivered as enema (and repeated once in the subgroup of patients with C. dif. infection) of 350 ml of standardised mixed transplantate prepared from faeces of 7 healthy donors.

Control group: Standard-of-care protocolised treatment of postantibiotic diarhea (which includes vancomycine 250 mg p.o. 6 hourly in the subgroup with C. dif. infection).

Primary outcome: Percentage of patients with treatment failure at day 7 after randomisation, which is defined as treatment either not being delivered or not being effective.

Secondary and exploratory outcomes: Influence of the intervention on colonic microbiome and metabolome, small bowel and colonic permeability, bacterial translocation and systemic inflammation response to procedure.

ELIGIBILITY:
Inclusion Criteria:

* signing of informed consent (see below)
* age > 18 yrs.
* in-patient in ICU or HDU (incl. burn unit) and expected to stay for >7 days
* diarrhea following antibiotic treatment defined as 3 or more stools per day or Bristol type 7 stool in the volume >300 ml/day if stool derivative device is in place, persisting for 24 hours despite enteral feeding formula has been stopped.

Exclusion Criteria:

* death appears imminent or ceilings of care put in place
* presence of new-onset sepsis defined as per 2016 definition
* lactate >2.0 mM, colon diameter > 9 cm on plain AXR
* the necessity of ongoing antibiotic treatment for another reasons
* unable to tolerate enema for any reason (e.g. surgery of the GI tract in the past year)
* pregnant and lactating woman
* patients with a history of severe anaphylactic food allergy, any other reason which - as per judgement of the treating clinician - makes faecal transplantation unsafe or not feasible (Note: All screening failures based on this criterion will be reported separately, inc. the reason why it was considered unsafe or not feasible to proceed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 7 days after randomisation
  Difference of proportion of patients between intervention and control groups in whom the treatment failed. Failure is defined as treatment has either not been delivered or has not been effective to cure diarrhoea as per WHO definition

SECONDARY OUTCOMES:
Comparison of therapeutic efficacy | 7 days after randomisation
  Difference of proportion of patients between intervention and control groups who are diarhoea-free (WHO definition)
Systemic inflammation | 7 days after randomisation
  Difference between intervention and control group in area under C-reactive protein plasma concentration curve
Organ failures | 7 days after randomisation
  Difference between intervention and control group in SOFA score curve
Postprocedural bacteriaemia | 3 hours after intervention
  Difference between intervention and control group in the percentage of positive blood cultures
Mortality | 28 day or hospital discharge, whichever occurs earlier
  Difference between intervention and control group in the absolute risk of death (intention-to-treat analysis)

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Kralovske Vinohrady University Hospital, Prague
  - František Duška, Prague, Česká Republika

REFERENCES:
- [Derived] Cibulkova I, Rehorova V, Soukupova H, Waldauf P, Cahova M, Manak J, Matejovic M, Duska F. Allogenic faecal microbiota transplantation for antibiotic-associated diarrhoea in critically ill patients (FEBATRICE)-Study protocol for a multi-centre randomised controlled trial (phase II). PLoS One. 2024 Dec 27;19(12):e0310180. doi: 10.1371/journal.pone.0310180. eCollection 2024. PMID 39729440

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT05430269/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT05430269/ICF_001.pdf